CLINICAL TRIAL: NCT06450808
Title: Die Mikroalge Phaeodactylum Tricornutum Ein Potentieller Fischersatz?- Pharmakokinetische Studie
Brief Title: The Microalga Phaeodactylum Tricornutum a Potential Fish Substitute?- Pharmacokinetic Study
Acronym: MikroFisch
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MikroFisch
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Pharmacokinetic Parameters

STUDY DESIGN:
Intervention Model Description: This study is a prospective blinded intervention study in a cross-over design with three single-dose treatment periods (2 %, 3 % and 4 % PT content in the investigational product) and a 14-day washout phase between the treatment periods.
Who Masked: Care Provider
Masking Description: Crossover: Three single-dose treatment periods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pesto with 3% Phaeodactylum (Experimental): Dried Microalgae integrated in the Pesto
  Interventions: Dietary Supplement: Dried Microalgae biomass
- Pesto with 4% Phaeodactylum (Experimental): Dried Microalgae integrated in the Pesto
  Interventions: Dietary Supplement: Dried Microalgae biomass
- Pesto with 5% Phaeodactylum (Experimental): Dried Microalgae integrated in the Pesto
  Interventions: Dietary Supplement: Dried Microalgae biomass

INTERVENTIONS:
Dietary Supplement: Dried Microalgae biomass — The products to be tested are pestos enriched with different amounts of the microalgae Phaeodactylum tricornutum (3, 4 and 5%). After drying, the microalgae Phaeodactylum, which has already been used in two previous applications (application german ethic F-2020-001), is added to the pesto. Three different pestos will be produced and enriched with different amounts of the microalgae Phaeodactylum.

SUMMARY:
In a cross-over design, pestos enriched with different levels of the microalgae Phaeodactylumtricornutum (2-3-4%) will be tested. The bioavailability of long-chain omega-3 fatty acids, in particular EPA and carotenoids, will be analysed in blood plasma postprandially within two days after a single dose. Pharmacokinetic parameters will be calculated from the measured data. The aim of the study is to gain insight into the bioavailability of selected microalgae constituents and the acceptance of microalgae pesto.

DETAILED DESCRIPTION:
The main objective of the project "Healthy nutrition through microalgae as a fish substitute" with the acronym MikroFisch, is to develop a novel fish substitute product based on microalgae biomass that provides us with essential nutrients. More and more people are interested in a healthy, sustainable diet and are looking for plant-based alternatives. These are available in a wide variety for meat, but not for fish, although sources of essential nutrients such as eicosapentaenoic acid and docosahexaenoic acid are urgently needed, which is where our concept of evaluating microalgae as a future food comes in. Based on current trends, the investigators see great development potential for our approach. The prerequisites for this are proof of the non-toxicity of the microalgae used, sufficient absorption of the nutrients they contain in the human gut, and the development of a presentation form that is suitable for food technology and sensory analysis. If these requirements can be met, a food product based on microalgae could enjoy a high level of acceptance. The Institute of Nutritional Medicine at the University of Hohenheim has been researching the microalgae PT for several years. As PT is not authorised as a novel food, studies on the suitability of the microalgae as a foodstuff must be carried out. The aim of the study is to characterise the pharmacokinetics of the dried microalgae Phaeodactylum tricornutum processed in a pesto ("investigational product") in healthy volunteers/patients in order to gain insights into its absorption, distribution in the organism, metabolisation and excretion. In particular, the time courses of the plasma concentrations of eicosapentaenoic acid (EPA) and the carotenoids fucoxanthin and b-carotene will be analysed, and the microalgae must also be properly processed into a tasty product before it can be used as food. For this reason, the concentration-dependent acceptance of the dosage form of the microalgae is also being analysed.

ELIGIBILITY:
Inclusion Criteria:

* Good general condition (investigator's decision)
* Declaration of consent for participation in the study

Exclusion Criteria:

* Acute illnesses or infectious diseases of any kind
* Chronic diseases that could influence the study results (investigator's decision)
* Chronic intestinal diseases and gastritis are exclusion criteria other than than CHD / COPD / neuromuscular diseases
* Known allergies to algae or Algae or pesto components
* smokers
* Pregnancy/breastfeeding period (anamnestic survey)
* Withdrawal of consent or lack of written consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC)- Eicosapentaonic acid | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Area under the curve (AUC)- Fucoxanthin | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Area under the curve (AUC)- B-Carotin | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Maximum Plasma Concentration [Cmax] of Eicosapentaonic acid | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Maximum Plasma Concentration [Cmax] of Fucoxanthin | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Maximum Plasma Concentration [Cmax] of B-Carotin | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Time of the maximum measured plasma concentration (max) of Eicosapentaonic acid | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Time of the maximum measured plasma concentration (max) of Fucoxanthin | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma
Time of the maximum measured plasma concentration (max) of B--Carotin | zero to 48 hours, during the whole study
  pharmacokinetic parameters measured in blood plasma

SECONDARY OUTCOMES:
Acceptance index of the pesto | 3 times of each pesto dose were Testet (the Microalgae is added zu 3%, 4% and 5% to the Pesto)
  A scale of 1 to 9 was used in this tasting study, labelled: 1=I don't like it at all; 5=neither; 9=I really like it. The categories to be evaluated were colour, smell, taste, texture and general acceptability.
Diagnostic markers in the blood | 4 times (at the Screening, At the study period 1, at the study period 2 and 3)
  Laboratory parameters
Omega-3/ Omega-6 ratio | 28 times (at the Screening, At the study period 1 (9 x), at the study period 2 (9x) and period 3 (9x), One period means before eating the pesto Timepoint 0, after 1h, after 2h, 4h, 6h,8h,10h,24h,48h
  in plasma measurement
Evaluation of the food diary, MEDAS questionnaire, FFQ questionnaire | the food diary is kept 3 x during the 3-day study, the MEDAS and FFQ are filled out once at the beginning of the study
  questionnaire to document food intake

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided